CLINICAL TRIAL: NCT04560972
Title: A Phase Ib Open-Label Study of LB-100 in Combination With Carboplatin/Etoposide/Atezolizumab in Untreated Extensive-Stage Small Cell Lung Carcinoma
Brief Title: LB-100, Carboplatin, Etoposide, and Atezolizumab for the Treatment of Untreated Extensive-Stage Small Cell Lung Cancer
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: City of Hope Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20068; NCI-2020-04297 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 20068 (Other: City of Hope Comprehensive Cancer Center); P30CA033572 (NIH)
Record Dates: First submitted 2020-06-22; First posted 2020-09-23 (Actual); Last update posted 2025-11-10 (Actual); Status verified 2025-11

CONDITIONS: Extensive Stage Lung Small Cell Carcinoma
MeSH Terms: interventions — atezolizumab; Carboplatin; Etoposide; LB100

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment (LB-100, carboplatin, etoposide, atezolizumab) (Experimental): INDUCTION: Patients receive LB-100 IV over 15 minutes on days 1 and 3, atezolizumab IV over 30-60 minutes on day 1, carboplatin IV over 30-60 minutes on day 1, and etoposide IV over 60 minutes on days 1-3. Treatment repeats every 21 days for 4 cycles in the absence of disease progression or unacceptable toxicity.
  MAINTENANCE: After completion of induction therapy, patients receive LB-100 IV over 15 minutes on days 1 and 3 and atezolizumab IV over 30 minutes on day 1. Cycles repeat every 21 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Atezolizumab; Drug: Carboplatin; Drug: Etoposide; Drug: Protein Phosphatase 2A Inhibitor LB-100

INTERVENTIONS:
Drug: Atezolizumab — Given IV
  Other Names: MPDL 3280A; MPDL 328OA; MPDL-3280A; MPDL3280A; MPDL328OA; RG7446; RO5541267; Tecentriq
Drug: Carboplatin — Given IV
  Other Names: Blastocarb; Carboplat; Carboplatin Hexal; Carboplatino; Carboplatinum; Carbosin; Carbosol; Carbotec; CBDCA; Displata; Ercar; JM-8; Nealorin; Novoplatinum; Paraplatin; Paraplatin AQ; Paraplatine; Platinwas; Ribocarbo
Drug: Etoposide — Given IV
  Other Names: Demethyl Epipodophyllotoxin Ethylidine Glucoside; EPEG; Lastet; Toposar; Vepesid; VP 16; VP 16-213; VP-16; VP-16-213; VP16
Drug: Protein Phosphatase 2A Inhibitor LB-100 — Given IV
  Other Names: LB-100; PP2A Inhibitor LB-100

SUMMARY:
This phase Ib trial studies the side effects and best dose of LB-100 when given together with carboplatin, etoposide, and atezolizumab for the treatment of untreated extensive-stage small cell lung cancer. Drugs such as carboplatin and etoposide work in different ways to stop the growth of tumor cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Immunotherapy with monoclonal antibodies, such as atezolizumab, may help the body's immune system attack the cancer, and may interfere with the ability of tumor cells to grow and spread. LB-100 has been shown to make anticancer drugs (chemotherapy) work better at killing cancer. LB-100 blocks a protein on the surface of cells called PP2A. Blocking this protein makes the tumor cells that express PP2A divide. This allows standard chemotherapy drugs such as carboplatin, etoposide, and atezolizumab work better at killing the tumor cells since these drugs work best at destroying cells that are dividing. Giving LB-100 in combination with standard chemotherapy drugs may work better to treat extensive-stage small cell lung cancer compared to standard chemotherapy drugs alone.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To determine the recommended phase II dose (RP2D) of protein phosphatase 2A inhibitor LB-100 (LB-100) when given in combination with standard carboplatin/etoposide/atezolizumab in treatment naive patients with extensive-stage small cell lung cancer (ED-SCLC).

SECONDARY OBJECTIVES:

I. To assess objective response rate (ORR). II. To assess progression-free survival (PFS). III. To assess overall survival (OS). IV. To assess duration of overall response (DOR). V. To assess safety and adverse events (AEs).

EXPLORATORY OBJECTIVES:

I. The pharmacokinetics (PK) of LB-100 and etoposide. II. The biomarkers relevant to LB-100 and the disease state as well as their correlation to clinical outcomes.

OUTLINE: This is a dose-escalation study of LB-100.

INDUCTION: Patients receive LB-100 intravenously (IV) over 15 minutes on days 1 and 3, atezolizumab IV over 30-60 minutes on day 1, carboplatin IV over 30-60 minutes on day 1, and etoposide IV over 60 minutes on days 1-3. Treatment repeats every 21 days for 4 cycles in the absence of disease progression or unacceptable toxicity.

MAINTENANCE: After completion of induction therapy, patients receive LB-100 IV over 15 minutes on days 1 and 3 and atezolizumab IV over 30 minutes on day 1. Cycles repeat every 21 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed for up to 30 days, and patients who discontinue study treatment without disease progression are followed every 6-8 weeks thereafter.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed extensive-stage disease small cell lung carcinoma per the Veterans Administration Lung Study Group (VALG) staging system
* Measurable disease as defined by Response Evaluation Criteria in Solid Tumors (RECIST): Revised RECIST guideline (version 1.1)
* Estimated life expectancy of at least 12 weeks
* For women: Must be surgically sterile (surgical procedure: bilateral tubal ligation), post-menopausal (at least 12 consecutive months of amenorrhea) or have a negative pregnancy test. Women of childbearing potential must be compliant with a medically approved contraceptive regimen (intrauterine device [IUD], birth control pills, or barrier device) during and for 3 months after the treatment period; must have a negative serum or urine pregnancy test within 14 days before study drug treatment and must not be breastfeeding
* For men: agreement to remain abstinent or use medically approved contraceptive measures, as defined below:

  * With female partners of childbearing potential or pregnant female partners, men must remain abstinent or use a condom during study therapy and for at least 6 months after the last dose of study therapy to avoid exposing the embryo
* A performance status of 0-2 on the Eastern Cooperative Oncology Group (ECOG) scale
* Absolute neutrophil (segmented and bands) count (ANC) >= 1.5 x 10/L
* Platelets >= 100 x 10/L
* Hemoglobin >= 9 g/dL
* Bilirubin =< 1.5 times upper limits of normal (ULN) may be enrolled
* Alkaline phosphatase (AP), alanine aminotransferase (ALT) and aspartate aminotransferase (AST) =< 3.0 times ULN (AP, AST, and ALT =< 5 times ULN are acceptable if the liver has tumor involvement)
* Calculated creatinine clearance (CrCl) >= 60 mL/min based on the Cockcroft and Gault formula
* All subjects must have the ability to understand and the willingness to sign a written informed consent
* No prior systemic chemotherapy, immunotherapy, biological, hormonal, or investigational therapy for SCLC

Exclusion Criteria:

* Currently enrolled in, or discontinued within the last 30 days from, a clinical trial involving an investigational product or non-approved use of a drug or device, or concurrently enrolled in any other type of medical research judged not to be scientifically or medically compatible with this study
* Diagnosis of non-small cell lung cancer (NSCLC) or mixed NSCLC and small cell lung cancer (SCLC)
* No prior malignancy other than SCLC, carcinoma in situ of the cervix, or nonmelanoma skin cancer, unless that prior malignancy was diagnosed and definitively treated 5 or more years prior to study entry with no subsequent evidence of recurrence. Patients with a history of low grade (Gleason score =< 6 = Gleason group 1) localized prostate cancer will be eligible even if diagnosed less than 5 years prior to study entry
* Serious concomitant systemic disorder that, in the opinion of the investigator, would compromise the patient's ability to adhere to the protocol
* Active or ongoing infection during screening requiring the use of systemic antibiotics
* Serious cardiac condition, such as myocardial infarction within 6 months, angina, or heart disease as defined by the New York Heart Association class III or IV
* Clinical evidence of central nervous system (CNS) metastases or leptomeningeal carcinomatosis, except for individuals who have previously-treated CNS metastases, are asymptomatic, and have had no requirement for steroid medication for 1 week prior to the first dose of study drug and have completed radiation 2 weeks prior to the first dose of study drug
* Known or suspected allergy to any agent given in association with this trial
* Pregnant or lactating women
* History of autoimmune disease, including minor/mild autoimmune disease not requiring immunosuppressants (such as eczema on less than 10% of the body surface area and long term diabetes mellitus type 1 on stable insulin)
* Known hepatitis B or hepatitis C
* Known human immunodeficiency virus (HIV) positive
* Treatment with systemic corticosteroid or other immunosuppressive medication. The use of inhaled corticosteroids for chronic obstructive pulmonary disease, mineralocorticoids (e.g., fludrocortisone) for patients with orthostatic hypotension, and low-dose supplemental corticosteroids for adrenocortical insufficiency are allowed
* Administration of a live, attenuated vaccine within 28 days prior to study
* Uncontrolled pleural effusion, pericardial effusion, or ascites requiring recurrent drainage procedures (once monthly or more frequently). Patients with indwelling catheters are allowed
* Uncontrolled or symptomatic hypercalcemia (> 1.5 mmol/L ionized calcium or calcium > 12 mg/dL or corrected serum calcium > ULN). Patients who are receiving denosumab prior to study entry must be willing and eligible to discontinue its use and replace it with a bisphosphonate while in the study
* History of idiopathic pulmonary fibrosis, organizing pneumonia (e.g., bronchiolitis obliterans), drug-induced pneumonitis, idiopathic pneumonitis, or evidence of active pneumonitis on screening chest computed tomography (CT) scan. History of radiation pneumonitis in the radiation field (fibrosis) is permitted
* Prior allogeneic bone marrow transplantation or solid organ transplant
* QTcF (Fridericia Correction Formula) > 470 on 2 out of 3 electrocardiograms (EKG's)
* Diagnosis of congenital long QT syndrome
* Treatment, within 7 days prior to first dose of study drug, with medications that are known to prolong the QT interval and/or are associated with a risk of torsades de pointes
* Treatment with CYP450 substrates within 7 days prior to first dose of study drug
* Treatment with nephrotoxic compounds within 7 days prior to first dose of study drug
* Treatment with warfarin within 7 days prior to first dose of study drug
* Treatment with antiepileptic medications that may increase etoposide clearance (including but not limited to phenytoin, phenobarbital, carbamazepine, and valproic acid) within 7 days prior to first dose of study drug
* Treatment with strong P-glycoprotein inhibitors within 7 days prior to first dose of study drug
* Subjects, who in the opinion of the investigator, may not be able to comply with the safety monitoring requirements of the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2021-05-28 (Actual); Primary Completion 2026-03-09 (Estimated); Study Completion 2026-03-09 (Estimated)

PRIMARY OUTCOMES:
Recommended phase II dose (RP2D) | End of first cycle (21 days)
  Measured using dose-limiting toxicity (DLT) during the first cycle as assessed by Common Terminology Criteria for Adverse Events (CTCAE) version 5.0.

SECONDARY OUTCOMES:
Objective response rate (ORR) | Up to 2 years
  Measured by Response Evaluation Criteria in Solid Tumors (RECIST) v1.1. Patients who respond to treatment and die without progressive disease (PD) (including death from study disease), duration of response will be censored at the date of the last objective progression-free disease assessment. For responding patients not known to have died as of the data cut-off date and who do not have PD, duration of response will be censored at the last progression-free assessment date. For responding patients who receive subsequent anticancer therapy (after discontinuation from all study treatment excluding PCI) prior to disease progression, duration of response will be censored at the date of last progression-free assessment prior to the initiation of post discontinuation anticancer therapy.
Duration of overall response | Up to 2 years
  Measured by RECIST v1.1.
Incidence of safety and adverse events | Up to 2 years
  Assessed by CTCAE version 5.0.
Progression-free survival (PFS) | Up to 2 years
  As defined by RECIST v1.1.
Overall survival (OS) | Time from the date of study enrollment to the date of death from any cause, assessed up to 2 years
  OS which is defined as the time from the date of study enrollment to the date of death from any cause. For patients who are still alive as of the data cutoff date, OS time will be censored on the date of the patient's last contact (last contact for patients in post discontinuation is last known alive date in mortality status).

OTHER OUTCOMES:
Cmax of LB-100 | Cycle 1 day 1: Pre-dose, immediately post LB-100 infusion, at 15 & 30 minutes, at 1, 2, 4, and 8 hours post LB-100 infusion (Each cycle is 21 days); Cycle 1, days 2-3: Pre-dose and 24 hours post LB-100 infusion (Each cycle is 21 days)]
  Plasma sampling for pharmacokinetic (PK) measurements of LB-100 will be performed . Blood samples will be collected to determine the Cmax of LB-100.
Cmax of endothall | Cycle 1 day 1: Pre-dose, immediately post LB-100 infusion, at 15 & 30 minutes, at 1, 2, 4, and 8 hours post LB-100 infusion (Each cycle is 21 days); Cycle 1, days 2-3: Pre-dose and 24 hours post LB-100 infusion (Each cycle is 21 days)]
  Plasma sampling for pharmacokinetic (PK) measurements of endothall, the metabolite of LB-100, will be performed .
  Blood samples will be collected to determine the Cmax of endothall.
Tmax of LB-100 | Cycle 1 day 1: Pre-dose, immediately post LB-100 infusion, at 15 & 30 minutes, at 1, 2, 4, and 8 hours post LB-100 infusion (Each cycle is 21 days); Cycle 1, days 2-3: Pre-dose and 24 hours post LB-100 infusion (Each cycle is 21 days)]
  Plasma sampling for pharmacokinetic (PK) measurements of LB-100 will be performed . Blood samples will be collected to determine the Tmax of LB-100.
Tmax of endothall | Cycle 1 day 1: Pre-dose, immediately post LB-100 infusion, at 15 & 30 minutes, at 1, 2, 4, and 8 hours post LB-100 infusion (Each cycle is 21 days); Cycle 1, days 2-3: Pre-dose and 24 hours post LB-100 infusion (Each cycle is 21 days)]
  Plasma sampling for pharmacokinetic (PK) measurements of endothall, the metabolite of LB-100, will be performed .
  Blood samples will be collected to determine the Tmax of endothall.
t1/2 of LB-100 | Cycle 1 day 1: Pre-dose, immediately post LB-100 infusion, at 15 & 30 minutes, at 1, 2, 4, and 8 hours post LB-100 infusion (Each cycle is 21 days); Cycle 1, days 2-3: Pre-dose and 24 hours post LB-100 infusion (Each cycle is 21 days)]
  Plasma sampling for pharmacokinetic (PK) measurements of LB-100 will be performed . Blood samples will be collected to determine the t1/2 of LB-100.
t1/2 of endothall | [Time Frame: Cycle 1 day 1: Pre-dose, immediately post LB-100 infusion, at 15 & 30 minutes, at 1, 2, 4, and 8 hours post LB-100 infusion (Each cycle is 21 days); Cycle 1, days 2-3: Pre-dose and 24 hours post LB-100 infusion (Each cycle is 21 days)]
  Plasma sampling for pharmacokinetic (PK) measurements of endothall, the metabolite of LB-100, will be performed .
  Blood samples will be collected to determine the t1/2 of endothall.
AUC0-t of LB-100 | Cycle 1 day 1: Pre-dose, immediately post LB-100 infusion, at 15 & 30 minutes, at 1, 2, 4, and 8 hours post LB-100 infusion (Each cycle is 21 days); Cycle 1, days 2-3: Pre-dose and 24 hours post LB-100 infusion (Each cycle is 21 days)]
  Plasma sampling for pharmacokinetic (PK) measurements of LB-100 will be performed . Blood samples will be collected to determine the AUC0-t of LB-100.
AUC0-t of endothall | Cycle 1 day 1: Pre-dose, immediately post LB-100 infusion, at 15 & 30 minutes, at 1, 2, 4, and 8 hours post LB-100 infusion (Each cycle is 21 days); Cycle 1, days 2-3: Pre-dose and 24 hours post LB-100 infusion (Each cycle is 21 days)]
  Plasma sampling for pharmacokinetic (PK) measurements of endothall, the metabolite of LB-100, will be performed .
  Blood samples will be collected to determine the AUC0-t of endothall.
CL of LB-100 | Cycle 1 day 1: Pre-dose, immediately post LB-100 infusion, at 15 & 30 minutes, at 1, 2, 4, and 8 hours post LB-100 infusion (Each cycle is 21 days); Cycle 1, days 2-3: Pre-dose and 24 hours post LB-100 infusion (Each cycle is 21 days)]
  Plasma sampling for pharmacokinetic (PK) measurements of LB-100 will be performed . Blood samples will be collected to determine the CL of LB-100.
CL of endothall | Cycle 1 day 1: Pre-dose, immediately post LB-100 infusion, at 15 & 30 minutes, at 1, 2, 4, and 8 hours post LB-100 infusion (Each cycle is 21 days); Cycle 1, days 2-3: Pre-dose and 24 hours post LB-100 infusion (Each cycle is 21 days)]
  Plasma sampling for pharmacokinetic (PK) measurements of endothall, the metabolite of LB-100, will be performed .
  Blood samples will be collected to determine the CL of endothall.
Relative abundance of immune cell populations | Up to 2 years]
  The signaling states that evolve in immune cells during treatment and that differentiate responders from nonresponders.
  Number of effector memory T cells Number of classical monocytes

CONTACTS AND LOCATIONS:
Overall Officials: Ravi Salgia, Principal Investigator — City of Hope Medical Center
Locations (1):
- City of Hope Medical Center, Duarte, California, United States

REFERENCES:
- [Derived] Feng Y, Massarelli E, Forman E, Kovach JS, Salgia R, Synold TW. An LC-MS/MS method for simultaneous determination of LB-100 and its active metabolite, endothall, in human plasma. Bioanalysis. 2023 Sep;15(17):1095-1107. doi: 10.4155/bio-2023-0078. Epub 2023 Aug 16. PMID 37584370